CLINICAL TRIAL: NCT02547480
Title: Pharmacokinetic Study In Patients With Liver Predominant Unresectable mCRC Receiving Treatment With LifePearl Microspheres Loaded With Irinotecan
Brief Title: LifePearl-Iri Pharmacokinetic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T126E2
Record Dates: First submitted 2015-08-27; First posted 2015-09-11 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Colorectal Cancer; mCRC
Keywords: liver; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TACE with irinotecan loaded LifePearl (Experimental): 10 patients receiving unilobar treatment: day 1=chemoembolization of first lobe of liver, day 14=chemoembolization of second lobe of liver, day 30=chemoembolization of first lobe of liver, day 44= chemoembolization of second lobe of liver; AND 10 patient receiving bilobar treatment: day 1=chemoembolization of both lobes of the liver, day 30=chemoembolization of both lobes of the liver
  Interventions: Device: TACE with irinotecan loaded LifePearl

INTERVENTIONS:
Device: TACE with irinotecan loaded LifePearl — Arterial embolization will be performed through lobar infusion and using a microcatheter. LifePearl microspheres of 200 µm will be used as preferred beads. They will be loaded with the appropriate dose of irinotecan hydrochloride injectable solution, mixed with the contrast media and distributed to the targeted lobe. The targeted dose is 100 mg of irinotecan per lobe treated, meaning that when treated unilobarly at baseline the total dose received will be 100 mg ( all in one lobe) and in during bilobar treatment, 200 mg in both lobes.
  Other Names: TACE

SUMMARY:
The primary purpose of the study is to evaluate the pharmacokinetic profile, safety, and efficacy of LifePearl microspheres loaded with irinotecan in the treatment of liver predominant mCRC by chemoembolization.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Histologically proven mCRC
* At least 1 measurable liver metastasis > 1 cm (mRECIST) Liver predominant disease ( ≥ 80% of metastatic disease confined to the liver)
* No portal vein involvement
* Performance status 0 or 1
* Life Expectancy ≥ 3m
* Adequate Hematologic function (ANC≥1.5 10^9/l; PLT≥75 10^9/l; INR (international normalized ratio) ≤1.3)
* Adequate liver and renal function (Total bilirubin ≤2.0 mg/dl; ALBUMINE 2.5g/dl; Serum creatinine ≤2.0 mg/dl; ALT (alanine transaminase),AST (aspartate transaminase) ≤5 times ULN)
* Less than 50% liver tumor replacement
* Patient has provided written informed consent
* Patient is affiliated to social security or equivalent system (France only)

Exclusion Criteria:

* Eligible for curative treatment (resection/RFA) History of hepaticocholangiojejunostomy or obstructive biliary disease (with/without previous treatment)
* Previous liver embolization
* Contraindication for intra-arterial embolization and local irinotecan administration
* Allergy to contrast media
* Patient is co-treated with potent CYP3A4/UGT1A1 (cytochrome P450 3A4/uridine diphosphate glucuronosyltransferase 1A1) inducers, i.e. rifampin, rifabutin, phenytoin, phenobarbital, carbamazepine and St John's Wort
* Patient is currently participating in a clinical trial with an investigational drug or a device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Patient is under judicial protection (France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04-28 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 2 days
  Maximum observed plasma concentrations of Irinotecan and its active metabolite SN38
Time to reach Cmax (Tmax) | 2 days
  Tmax will be estimated directly from concentration-time data
Area Under the Curve (AUC) | 1 day
  The trapezoidal rule will be used to calculate the area under the curve over 24 hours

SECONDARY OUTCOMES:
Adverse Events (AE) (grade ≥3) and Serious AEs related with study treatment up to 30 days post initial treatment | 1 month
Overall Survival | 12 months
Progression-Free Survival | 12 months
Response rate | 3 months
  Response rate (mRECIST criteria) 3 months after the first treatment
Technical success - treatment delivery | 1 day
  Ability to deliver ≥75% of the planned dose during the first chemoembolization
Technical success - total dose delivered | 6 weeks
  Sum of all doses delivered during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hans Prenen, MD, Principal Investigator — Universitair Ziekenhuis Leuven; Philippe Pereira, MD, Principal Investigator — SLK Kliniken Heilbronn GmbH; Julien Taieb, MD, Principal Investigator — Hôpital Georges Pompidou Paris
Locations (3):
- KUL, Leuven, Belgium
- Germany (2):
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Klinikum Bogenhausen, Städt. Klinikum München GmbH, Munich